CLINICAL TRIAL: NCT02781831
Title: Clinical Feasibility and Efficacy of Robot-assisted Gait Training for Improving Motor Functions in Patients With Stroke
Brief Title: Robot-assisted Gait Training for Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: HIWIN Technologies Corporation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIWIN-CMU-C-105-1
Record Dates: First submitted 2016-05-03; First posted 2016-05-25 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Rehabilitation (Active Comparator): Patient with stroke receiving standard hospital based rehabilitation program
  Interventions: Procedure: Standard rehab
- Robot-assisted Rehabilitation (Experimental): Patient with stroke receiving standard hospital based rehabilitation as well as robot-assisted gait rehabilitation program
  Interventions: Device: Robot-assisted gait rehabilitation

INTERVENTIONS:
Procedure: Standard rehab — Standard hospital based rehabilitation for patients with stroke
  Arms: Standard Rehabilitation
Device: Robot-assisted gait rehabilitation — An extra 30 minutes of robot-assisted gait rehabilitation after receiving standard hospital based rehabilitation for patients with stroke
  Arms: Robot-assisted Rehabilitation

SUMMARY:
Investigation of the clinical feasibility and efficacy of a newly developed robot-assisted gait training system for stroke survivors. It is anticipated that robot-assisted gait rehabilitation in combination with standard hospital based rehabilitation will achieve significantly better gait outcomes than standard hospital based rehabilitation alone.

DETAILED DESCRIPTION:
Stroke is the leading cause of permanent disability in most developed countries world wide with one-third of the surviving patients from stroke fail to regain independent walking ability. Robot-assisted gait rehabilitation that is able to deliver high intensity and consistent repeatability in a safe and controlled environment are gaining traction and advocators for its inclusion as part of the routine post-stroke rehabilitation program. However, despite the recent technological advances in the development and design of better robotics, the exact benefit of the robot-assisted therapy over traditional rehabilitation remain sparse and unclear. It is therefore the aim of the proposed project to fulfil this important gap in our clinical knowledge by comparatively investigate the clinical feasibility and efficacy of a recently developed HIWIN Robotic Gait Training System (MRG-P100) against the traditional rehabilitation program with an emphasis on the determination of functional recovery and the appropriate gait adaptation of such robotic system for stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Between the age of 20-65 years;
2. Diagnosis of first, single unilateral cortical-subcortical stroke verified by brain imaging;
3. Paresis of a lower limb;
4. Inability to walk without aid or device.

Exclusion Criteria:

1. Deemed by a physician to be medically unstable;
2. Other prior musculoskeletal conditions that affected gait capacity;
3. Co-existence of other neurological diseases;
4. Cognitive impairments that would impact on the safe participation in the study (MMSE<23) -

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment, lower extremity subscale | Assessing change from baseline after 1 month of intervention
  Lower limb function as measured by Fugl-Meyer Assessment, lower extremity subscale

SECONDARY OUTCOMES:
Functional Ambulation Categories | Assessing change from baseline after 1 month of intervention
  Categorizes patients according to basic motor skills necessary for functional ambulation
10 Meters Walking Test | Assessing change from baseline after 1 month of intervention
  Assesses walking speed in meters per second over a short duration
Berg Balance Scale | Assessing change from baseline after 1 month of intervention
  testing a participant's static and dynamic balance abilities
Timed Up and Go test | Assessing change from baseline after 1 month of intervention
  Assess a participant's mobility and requires both static and dynamic balance
Kinetic and Kinematic Gait Analysis | Assessing change from baseline after 1 month of intervention
  The temporo-spatial and kinematic gait parameters of the participants will be assessed using a Vicon Motion Analysis System with kinetic data collection through a force plate.

CONTACTS AND LOCATIONS:
Overall Officials: Nai-Hsin Meng, M.D., Principal Investigator — China Medical University, China Medical University Hospital
Locations (1):
- China Medical University Hospial, Taichung, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided